CLINICAL TRIAL: NCT02410824
Title: Bilateral Dispensing Clinical Trial of Stenfilcon A Against Etafilcon A for Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV-15-02
Record Dates: First submitted 2015-03-31; First posted 2015-04-08 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stenfilcon A toric lens (Experimental): Participants were randomized to wear stenfilcon A toric lens for one week during the cross over study.
  Interventions: Device: stenfilcon A toric lens
- etafilcon A toric lens (Active Comparator): Participants were randomized to wear etafilcon A toric lens for one week during the cross over study.
  Interventions: Device: etafilcon A toric lens

INTERVENTIONS:
Device: stenfilcon A toric lens — toric contact lens
  Arms: stenfilcon A toric lens
Device: etafilcon A toric lens — toric contact lens
  Arms: etafilcon A toric lens

SUMMARY:
Bilateral dispensing clinical trial of stenfilcon A against etafilcon A for astigmatism.

DETAILED DESCRIPTION:
CooperVision is evaluating the clinical performance of an FDA cleared silicone-hydrogel lens material stenfilcon A (test) compared to etafilcon A for Astigmatism lens (control) when worn on a daily wear basis over one (1) week in a randomized, bilateral, cross-over, dispensing study.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age for Canada and 18 years of age for the USA and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Is an adapted soft contact lens wearer;
* Requires a spherical contact lens prescription between -1.00 to -6.00 inclusive in each eye
* Has spectacle astigmatism: -0.50 to -1.50D (Diopter) cylinder (Axis: 90±20, 180±20 in both eyes);
* Willing to wear contact lens in both eyes for at least 8 hours per day, 7 days per week;
* Has manifest refraction visual acuities (VA) equal to or better than logMAR equivalent of 20/25 in each eye;
* To be eligible for lens dispensing, the subject must have VA of logMAR equivalent of 20/30 or better in each eye with the study lenses and the investigator must judge the fit as acceptable.

Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Has any known active* ocular disease and/or infection;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Is pregnant, lactating (by verbal confirmation at the screening visit);
* Is aphakic;
* Has undergone refractive error surgery

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng C Lin, OD PhD, Principal Investigator — UC Berkeley Clinical Research Center
Locations (2):
- Clinical Research Center, University of California, Berkeley, Berkeley, California, United States
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 subjects discontinued before lens randomization due to screen failure.
Groups:
- Stenfilcon A Toric Lens, Then Etafilcon A Toric Lens: Participants were randomized to wear stenfilcon A toric lens for one week, then cross over to the etafilcon A toric lens.
  stenfilcon A: toric contact lens
  etafilcon A: toric contact lens
- Etafilcon A Toric Lens, Then Stenfilcon A Toric Lens: Participants were randomized to wear etafilcon A toric lens for one week, then cross over to the stenfilcon A toric lens.
  etafilcon A: toric contact lens
  stenfilcon A: toric contact lens
Period: First Intervention (One Week)
Arm/Group | Stenfilcon A Toric Lens, Then Etafilcon A Toric Lens | Etafilcon A Toric Lens, Then Stenfilcon A Toric Lens
Started | 22 | 23
Completed | 22 | 22
Not Completed | 0 | 1
Not completed — Headache | 0 | 1
Period: Second Intervention (One Week)
Arm/Group | Stenfilcon A Toric Lens, Then Etafilcon A Toric Lens | Etafilcon A Toric Lens, Then Stenfilcon A Toric Lens
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Baseline Characteristics: Participants were randomized to wear stenfilcon A toric lens or etafilcon A toric lens bilaterally for one week, then cross over to the alternative pair.
Arm/Group | Overall Baseline Characteristics
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 10
Region of Enrollment [Number; unit: participants]
  Canada | 21
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Subjective ratings of lens performance for comfort assessed at baseline and 1 week. Comfort Scale 0-100, 0=extremely uncomfortable/cannot tolerate, 100=extremely comfortable/cannot be felt.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stenfilcon A Toric Lens: Participants were randomized to wear stenfilcon A toric lens for one week during the cross over study.
  stenfilcon A: toric contact lens
- Etafilcon A Toric Lens: Participants were randomized to wear etafilcon A toric lens for one week during the cross over study.
  etafilcon A: toric contact lens
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline | 88 (13) | 78 (18)
  1 week | 85 (14) | 77 (21)

2. Primary Outcome: Handling
Description: Subjective ratings of lens performance for handling assessed at baseline and 1 week. Handling Scale 0-100, 0=very difficult to handle, 100=very easy to handle.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline | 87 (12) | 81 (16)
  1 week | 87 (18) | 81 (23)

3. Primary Outcome: Vision
Description: Subjective ratings of lens performance for vision assessed at baseline and 1 week. Scale 0-100, 0=extremely poor vision all of the time, cannot function, 100=excellent.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline | 83 (16) | 78 (21)
  1 week | 86 (17) | 83 (17)

4. Primary Outcome: High Visual Acuity
Description: High illumination high contrast (HIHC) visual acuity for stenfilcon A toric lens and etafilcon A toric lens assessed at baseline and 1 week. Visual acuity is measured by logMAR.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Stenfilcon A Toric Lens: Participants were randomized to wear stenfilcon A toric lens for one week during the cross over study.
  stenfilcon A: toric lens contact lens
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
LogMAR
  Baseline | -0.10 (0.06) | -0.08 (0.06)
  1 week | -0.09 (0.07) | -0.09 (0.07)

5. Primary Outcome: Low Visual Acuity
Description: Low illumination high contrast (LIHC) visual acuity for stenfilcon A toric lens and etafilcon A toric lens assessed at baseline and 1 week. Visual acuity is measured by logMAR.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
LogMAR
  Baseline | -0.08 (0.06) | -0.07 (0.06)
  1 week | -0.07 (0.07) | -0.07 (0.07)

6. Primary Outcome: Lens Surface - Wettability
Description: Lens surface of wettability for stenfilcon A toric lens and etafilcon A toric lens assessed at baseline and 1 week. Scale 0-4, 0=severely reduced, 4=excellent wettability.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline | 3.2 (0.8) | 3.4 (0.5)
  1 week | 3.2 (0.7) | 3.3 (0.7)

7. Primary Outcome: Lens Surface - Deposits
Description: Lens surface of wettability for stenfilcon A toric lens and etafilcon A toric lens assessed at baseline and 1 week. Scale 0-4, 0=no deposits, 4=severe deposits.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline | 0.09 (0.23) | 0.11 (0.24)
  1 week | 0.18 (0.28) | 0.25 (0.37)

8. Primary Outcome: Corneal Staining, Type
Description: Ocular health of corneal staining, type for stenfilcon A toric lens and etafilcon A toric lens assessed at baseline and 1 week. Scale 0-4, 0=No staining, 4=Severe staining Five quadrants: C - Central, N - Nasal, T - Temporal, S - Superior, I - Inferior
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline - Central | 0.09 (0.32) | 0.09 (0.32)
  1 week - Central | 0.07 (0.27) | 0.02 (0.21)
  Baseline - Nasal | 0.19 (0.42) | 0.19 (0.42)
  1 week - Nasal | 0.13 (0.54) | 0.22 (0.62)
  Baseline - Temporal | 0.09 (0.28) | 0.09 (0.28)
  1 week - Temporal | 0.01 (0.2) | 0.14 (0.42)
  Baseline - Superior | 0.12 (0.34) | 0.12 (0.34)
  1 week - Superior | 0.36 (0.62) | 0.24 (0.49)
  Baseline - Inferior | 0.56 (0.75) | 0.56 (0.75)
  1 week - Inferior | 0.30 (0.58) | 0.49 (0.79)

9. Primary Outcome: Corneal Staining, Extent
Description: Ocular health of corneal staining (extent) for stenfilcon A toric lens and etafilcon A toric lens assessed at baseline and 1 week. Scale 0-4, 0=No staining 1=1-15% of area 2=16-30% of area 3=31-45% of area 4=>45% of area Five quadrants: C - Central, N - Nasal, T - Temporal, S - Superior, I - Inferior
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline - Central | 0.07 (0.30) | 0.07 (0.30)
  1 week - Central | 0.07 (0.26) | 0.01 (0.11)
  Baseline - Nasal | 0.13 (0.30) | 0.13 (0.30)
  1 week - Nasal | 0.06 (0.25) | 0.14 (0.36)
  Baseline - Temporal | 0.09 (0.28) | 0.09 (0.28)
  1 week - Temporal | 0.02 (0.12) | 0.13 (0.38)
  Baseline - Superior | 0.09 (0.27) | 0.09 (0.27)
  1 week - Superior | 0.22 (0.46) | 0.20 (0.42)
  Baseline - Inferior | 0.47 (0.59) | 0.47 (0.59)
  1 week - Inferior | 0.28 (0.55) | 0.41 (0.61)

10. Primary Outcome: Conjunctival Staining
Description: Ocular health of conjunctival staining for stenfilcon A toric lens and etafilcon A toric lens assessed at baseline and 1 week. Measured in 0.50 steps, scale 0-4, 0=None, 1=Minimal diffuse punctate, 2=Coalescent punctate, 3=Confluent, 4= Deep confluent
  N - Nasal, T - Temporal, S - Superior, I - Inferior
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline - Nasal | 0.36 (0.60) | 0.36 (0.60)
  1 week - Nasal | 1.19 (0.82) | 1.49 (0.96)
  Baseline - Temporal | 0.28 (0.41) | 0.28 (0.41)
  1 week - Temporal | 1.06 (0.70) | 0.91 (0.76)
  Baseline - Superior | 0.09 (0.30) | 0.09 (0.30)
  1 week - Superior | 0.13 (0.34) | 0.09 (0.27)
  Baseline - Inferior | 0.22 (0.41) | 0.22 (0.41)
  1 week - Inferior | 0.68 (0.79) | 0.78 (0.96)

11. Primary Outcome: Lens Durability
Description: Lens durability (lens tearing) between stenfilcon A toric lens or etafilcon A toric lens assessed at 1 week. (The number of lens tear or lens nicks found during the one week study).
Time Frame: 1 Week
Measure: Number; unit: Lens tear or nick
Units Other Than Participants: Lenses
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
Number analyzed (Lenses) | 88 | 88
Lens tear or nick | 1 | 0

12. Primary Outcome: Lens Fit Acceptance
Description: Lens fit acceptance (on eye stability) for stenfilcon A and etafilcon A assessed at baseline and 1 week. Scale 0-4, 0=Can't be worn, 1=Poor, 2=Fair, 3=Good, 4=optimum.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline | 3.5 (0.3) | 3.4 (0.3)
  1 week | 3.5 (0.4) | 3.3 (0.4)

13. Secondary Outcome: Dryness
Description: Subjective ratings of lens performance for dryness assessed during the day and at the end of the day. Scale 0-100, 0=cannot be worn, extremely dry, 100=no dryness experienced at any time.
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  During the Day | 82 (18) | 74 (23)
  End of Day | 76 (21) | 67 (24)

14. Secondary Outcome: Overall Satisfaction
Description: Overall satisfaction of stenfilcon A and etafilcon A lenses. Scale 0-100, 0=extremely dissatisfied, 100=extremely satisfied.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline | 87 (13) | 80 (16)
  1 week | 83 (17) | 77 (23)

ADVERSE EVENTS:
Arm/Group | Stenfilcon A Toric Lens | Etafilcon A Toric Lens
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other